CLINICAL TRIAL: NCT02313207
Title: Confocal Endomicroscopy for the Detection of Food Intolerances in Patients With IBS.
Brief Title: Confocal Laser Endomicroscopy in IBS Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No appropriate participants
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Mark Ellrichmann, Senior Consultant, Unit of Experimental Endoscopy, University Hospital Schleswig-Holstein
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE-IBS-2
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: IBS; Food Intolerance
MeSH Terms: conditions — Food Intolerance | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FODMAP diet (Active Comparator): FODMAP diet for 2 weeks, patients will undergo a specific FODMAP diet for a period of 2 weeks.
  Interventions: Dietary Supplement: FODMAP
- Specific bread diet (Active Comparator): Specific bread diet eliminating wheat and yeast for 2 weeks, patients will undergo a specific FODMAP diet for a period of 2 weeks.
  Interventions: Dietary Supplement: FODMAP

INTERVENTIONS:
Dietary Supplement: FODMAP — patients will undergo a specific FODMAP diet for a period of 2 weeks.

SUMMARY:
This study will assess dynamic effects of two major antigens on the duodenal mucosa by confocal laser endomicroscopy (CLE). Patients will be blinded to the antigens used (wheat, yeast). Following CLE it is planned to have a cross over exclusion diet with/without the antigens including a washout phase. Furthermore, patients will undergo a 2 week FODMAP diet to be able to compare results found of both diets and allow to understand whether our findings of food intolerance will be better and more precise than a common FODMAP diet.

Post CLE food challenge patients biopsies will be taken for histology. They will then be randomized into two groups and blinded to the diet they undergo. They will be provided with a supply of custom-made bread they will have for 2 weeks (custom made by a bakery in Kiel). For one study arm bread will contain either wheat and yeast, for the other arm the bread will not contain these ingredients. The taste of the "normal" bread will be denaturised. Crossover will take place after a two-week washout phase.

ELIGIBILITY:
Inclusion Criteria:

IBS according to the Rome III criteria moderate/severe refractory daily symptoms >1year (FGID-C1) sub classified as IBS-D, constipation predominant (IBS-C) or mixed type (IBS-M) no past infection to trigger symptom no structural/ biochemical cause of their symptoms identified negative gastroscopy, colonoscopy including histology Worsening symptoms after meals various exclusion diets - ineffective females not menstruating during CLE no known allergy to methylene blue or fluorescein Age >18 years Negative routine testing for food intolerance (or known lactose/fructose intolerance) Positive informed consent

Exclusion Criteria:

no consent known reason for the abdominal pain and bloating other than lactose/fructose intolerance M. Whipple Known infectious gastrointestinal disease Stricture in the upper gastrointestinal tract Age <18years Impaired renal function (Creatinine >1.2 mg/dL) Pregnancy or breast-feeding Inability to obtain informed consent Active GI Bleeding Known allergy to Methylene blue or Fluorescein Participation in other clinical trials within the last 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Detection of mucosal reaction on allergen exposure | up to 5 sec

CONTACTS AND LOCATIONS:
Overall Officials: Annette Fritscher-Ravens, MD, PhD, Principal Investigator — University Hospital Schleswig-Holstein; Mark Ellrichmann, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig Holstein, Campus Kiel, Unit Experimental Endoscopy, Kiel, Germany